CLINICAL TRIAL: NCT05516498
Title: A Two Part Phase IIa/b Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Dose-ranging Study to Assess Efficacy, Safety, and Tolerability of the Combination of Zibotentan and Dapagliflozin, and Dapagliflozin Monotherapy Versus Placebo in Participants With Cirrhosis With Features of Portal Hypertension
Brief Title: Zibotentan and Dapagliflozin Combination, EvAluated in Liver Cirrhosis (ZEAL Study)
Acronym: ZEAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was ended earlier than planned due to a sponsor decision.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: D4326C00003; 2021-006577-30 (EudraCT Number)
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Treatment Group 1 (Experimental): Participants will receive once daily dose of placebo matching zibotentan capsule + placebo matching dapagliflozin tablet for 6 weeks.
  Interventions: Drug: Part A: Placebo (matching zibotentan capsule & matching dapagliflozin tablet)
- Part A: Treatment Group 2 (Experimental): Participants will receive once daily dose of zibotentan capsule + dapagliflozin tablet for 6 weeks.
  Interventions: Drug: Part A: zibotentan (dose B) + dapagliflozin
- Part B: Treatment Group 1 (Experimental): Participants will receive once daily dose of placebo matching zibotentan capsule + placebo matching dapagliflozin tablet for 16 weeks.
  Interventions: Drug: Part B: Placebo (matching zibotentan capsule & matching dapagliflozin tablet)
- Part B: Treatment Group 2 (Experimental): Participants will receive once daily dose of placebo matching zibotentan capsule + dapagliflozin tablet for 16 weeks.
  Interventions: Drug: Part B: placebo (matching zibotentan capsule) + dapagliflozin
- Part B: Treatment Group 3 (Experimental): Participants will receive once daily dose of zibotentan capsule + dapagliflozin tablet for 16 weeks.
  Interventions: Drug: Part B: zibotentan (dose A) + dapagliflozin
- Part B: Treatment Group 4 (Experimental): Participants will receive once daily dose of zibotentan capsule + dapagliflozin tablet for 16 weeks.
  Interventions: Drug: Part B: zibotentan (dose B) + dapagliflozin
- Part B: Treatment Group 5 (Experimental): Participants will receive once daily dose of zibotentan capsule + dapagliflozin tablet for 16 weeks.
  Interventions: Drug: Part B: zibotentan (dose C) + dapagliflozin

INTERVENTIONS:
Drug: Part A: Placebo (matching zibotentan capsule & matching dapagliflozin tablet) — placebo capsule (matching zibotentan capsule)
  placebo tablet (matching dapagliflozin tablet)
  Arms: Part A: Treatment Group 1
Drug: Part A: zibotentan (dose B) + dapagliflozin — zibotentan capsule
  dapagliflozin tablet
  Arms: Part A: Treatment Group 2
Drug: Part B: Placebo (matching zibotentan capsule & matching dapagliflozin tablet) — placebo capsule (matching zibotentan capsule)
  placebo tablet (matching dapagliflozin tablet)
  Arms: Part B: Treatment Group 1
Drug: Part B: placebo (matching zibotentan capsule) + dapagliflozin — placebo capsule (matching zibotentan capsule)
  dapagliflozin tablet
  Arms: Part B: Treatment Group 2
Drug: Part B: zibotentan (dose A) + dapagliflozin — zibotentan capsule
  dapagliflozin tablet
  Arms: Part B: Treatment Group 3
Drug: Part B: zibotentan (dose B) + dapagliflozin — zibotentan capsule
  dapagliflozin tablet
  Arms: Part B: Treatment Group 4
Drug: Part B: zibotentan (dose C) + dapagliflozin — zibotentan capsule
  dapagliflozin tablet
  Arms: Part B: Treatment Group 5

SUMMARY:
This is a two part Phase IIa/b multicentre, randomised, double-blind, placebo-controlled, parallel group dose-ranging study to assess the efficacy, safety, and tolerability of the combination of zibotentan and dapagliflozin, and dapagliflozin monotherapy versus placebo in participants with cirrhosis with features of portal hypertension.

DETAILED DESCRIPTION:
Part A will assess the efficacy, safety, and tolerability of the combination of B mg zibotentan and 10 mg dapagliflozin versus placebo in participants with Child-Pugh A cirrhosis with features of portal hypertension and with no history of decompensation events.

If the safety profile is determined to be acceptable at the conclusion of Part A, Part B will investigate efficacy, safety, and tolerability of A mg, B mg, or C mg zibotentan combined with 10 mg dapagliflozin and of 10 mg dapagliflozin monotherapy versus placebo in participants with cirrhosis with features of portal hypertension. Part B will include a broader range of Child- Pugh A and Child-Pugh B cirrhosis participants, including those with more severe disease, a history of decompensation events, or current ascites.

The study will be conducted in approximately 30 to 45 study centres in North America, Asia, and Europe.

ELIGIBILITY:
Study principal inclusion criteria For both Part A and Part B

1. No current or prior (within 1 month of enrolment) medical treatment with an SGLT2 inhibitor or ERAs.
2. On no or a stable dose of beta blockers, with no major dose changes within 1 month prior to the first dose of study intervention.
3. Provision of signed and dated, written ICF prior to any mandatory study-specific procedures, sampling, and analyses.
4. Female participants of non-childbearing potential confirmed at screening by fulfilling one of the following criteria:

   1. Post-menopausal: defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments; and also, FSH levels in the post-menopausal range by central laboratory.
   2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
5. Female participants must have a negative pregnancy test at screening and must not be lactating

Part A participants who have the following:

1. Clinical and/or histological diagnosis of cirrhosis with either (i) features of portal hypertension or (ii) liver stiffness ≥ 21 kPa.
2. MELD score < 15.
3. Child-Pugh score ≤ 6.
4. No clinically evident ascites.
5. No evidence of worsening of hepatic function (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status) within the last month prior to dosing, as determined by the investigator or usual practitioner.
6. HVPG recording of good enough quality as judged by a central reader.

Part B participants who have the following:

1. Clinical and/or histological diagnosis of cirrhosis and either history of decompensation or compensated cirrhosis with signs of clinically significant portal hypertension.
2. HVPG recording of good enough quality and HVPG > 10 mmHg, as judged by a central reader.
3. MELD score < 15.
4. Child-Pugh score < 10.
5. No ascites or ascites up to grade 2 without change in diuretic treatment within the last month prior to first dose and no paracentesis within the last month or planned paracentesis in the next 4 months at screening.
6. No evidence of worsening of hepatic function (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status) within the last month prior to dosing, as determined by the investigator or usual practitioner.

Study principal exclusion criteria:

1. Any evidence of a clinically significant disease which in the investigator's opinion makes it undesirable for the participant to participate in the study.
2. Liver cirrhosis caused by chronic cholestatic liver disease
3. ALT or AST ≥ 150 U/L and/or total bilirubin ≥ 3 × ULN
4. Acute liver injury caused by drug toxicity or by an infection.
5. Any history of hepatocellular carcinoma.
6. Liver transplant or expected liver transplantation within 6 months of screening.
7. History of TIPS or a planned TIPS within 6 months from enrolment into the study.
8. Active treatment for HCV within the last 1 year or HBV antiviral therapy for less than 1 year.
9. Participants with T1DM.

Medical Conditions (Part A only)

1. INR > 1.5.
2. Serum/plasma levels of albumin ≤ 35 g/L.
3. Platelet count < 75 × 109/L.
4. History of ascites
5. History of hepatic hydrothorax
6. History of portopulmonary syndrome
7. History of hepatic encephalopathy
8. History of variceal haemorrhage
9. History of acute kidney injury
10. History of heart failure, including high output heart failure (eg, due to hyperthyroidism or Paget's disease)

Medical Conditions (Part B only)

1. INR > 1.7.
2. Serum/plasma levels of albumin ≤ 28 g/L.
3. Platelet count < 50 × /109L.
4. Acute kidney injury within 3 months of screening.
5. History of encephalopathy of West Haven grade 2 or higher within 6 months prior to screening.
6. History of variceal haemorrhage within 6 months prior to screening.
7. NYHA functional heart failure class III or IV or with unstable heart failure requiring hospitalisation for optimisation of heart failure treatment and who are not yet stable on heart failure therapy within 6 months prior to screening.
8. Heart failure due to cardiomyopathies that would primarily require specific other treatment: eg, cardiomyopathy due to pericardial disease, amyloidosis or other infiltrative diseases, cardiomyopathy related to congenital heart disease, primary hypertrophic cardiomyopathy, cardiomyopathy related to toxic or infective conditions (ie, chemotherapy, infective myocarditis, septic cardiomyopathy).
9. High output heart failure (eg, due to hyperthyroidism or Paget's disease).
10. Heart failure due to primary cardiac valvular disease/dysfunction, severe functional mitral or tricuspid valve insufficiency, or planned cardiac valve repair/replacement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Part A: Absolute change in HVPG from baseline to Week 6. | at Week 6
  To evaluate the change from baseline in HVPG on zibotentan and dapagliflozin in combination versus placebo.
Part B: Absolute change in HVPG from baseline to Week 6. | at Week 6
  To evaluate the change from baseline in HVPG on zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo.

SECONDARY OUTCOMES:
Part A: Percent change in HVPG from baseline to Week 6. | at Week 6
  To evaluate the change from baseline in HVPG on zibotentan and dapagliflozin in combination versus placebo.
Part A: HVPG response, where a responder is defined as HVPG < 10 mmHg or a reduction in HVPG of ≥ 1.5 mmHg from baseline to Week 6. | at Week 6
  To evaluate the proportion of participants achieving HVPG < 10 mmHg or a reduction in HVPG of ≥ 1.5 mmHg on zibotentan and dapagliflozin versus placebo.
Part A: Evaluation of change in body weight (kg) over time course of study. Percentage and absolute change from baseline in body weight at Week 6. | at Week 6
  To evaluate the effect of zibotentan and dapagliflozin in combination versus placebo on change in body weight.
Part A: Percentage and absolute change in total dosage of loop-diuretic equivalents use from baseline to Week 6. | at Week 6
  To evaluate the effect of zibotentan and dapagliflozin in combination versus placebo on total loop-diuretic equivalents use.
Part A: Change in total body water, extracellular water and intracellular water volumes from baseline to Week 6. Change in total body fat mass from baseline to Week 6. | at Week 6
  To evaluate the effect of zibotentan and dapagliflozin in combination versus placebo on body water volumes and body fat mass.
Part A: Change in systolic and diastolic blood pressure from baseline to Week 6. | at Week 6
  To evaluate the effect of zibotentan and dapagliflozin in combination versus placebo on changes in office-based systolic and diastolic blood pressure.
Part B: Percentage change in HVPG from baseline to Week 6. | at Week 6
  To evaluate the change from baseline in HVPG on zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo.
Part B: HVPG response, where a responder is defined as at least 20% decrease or a reduction to or below 12 mmHg in HVPG from baseline to Week 6. | at Week 6
  To evaluate the proportion of participants achieving at least 20% decrease in HVPG or a reduction to or below 12 mmHg in HVPG on zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo.
Part B: Evaluation of change in body weight (kg) over time course of study. Percentage and absolute change from baseline in body weight at Week 6 and Week 16. | at Week 6 and Week 16
  To evaluate the effect of zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo on change in body weight.
Part B: Absolute change in total dosage of loop-diuretic equivalents use from baseline to Week 6 and Week 16. | at Week 6 and Week 16
  To evaluate the effect of zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo on total loop-diuretic equivalents use.
Part B: Change in total body water, extracellular water and intracellular water volumes from baseline to Week 6 and Week 16. Change in total body fat mass from baseline to Week 6 and Week 16. | at Week 6 and Week 16
  To evaluate the effect of zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo on body water volumes and body fat mass.
Part B: Change in systolic and diastolic blood pressure from baseline to Week 6 and Week 16. | at Week 6 and Week 16
  To evaluate the effect of zibotentan and dapagliflozin in combination and dapagliflozin monotherapy versus placebo on changes in office-based systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (11):
  - Research Site, Birmingham, Alabama
  - Research Site, Pasadena, California
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, Rochester, Minnesota
  - Research Site, The Bronx, New York
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Milwaukee, Wisconsin
- Research Site, Heidelberg, Australia
- Research Site, Vienna, Austria
- Research Site, Edegem, Belgium
- China (4):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
- Research Site, Prague, Czechia
- Denmark (4):
  - Research Site, Aarhus N
  - Research Site, Esbjerg
  - Research Site, Hvidovre
  - Research Site, Køge
- France (4):
  - Research Site, Angers
  - Research Site, Clichy
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Dresden
  - Research Site, Landshut
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Wiesbaden
- Research Site, Amsterdam, Netherlands
- Research Site, Cluj-Napoca, Romania
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Santander
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Lucerne
  - Research Site, Lugano
- Research Site, Taipei, Taiwan
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home